CLINICAL TRIAL: NCT05947149
Title: Health Related Quality of Life (HRQoL) in Patients With Solid Tumors Treated With Hadrontherapy (HadroQoL).
Brief Title: HRQoL in Patients With Solid Tumors Treated With Hadrontherapy
Acronym: HadroQoL
Status: Recruiting | Type: Observational
Sponsor: CNAO National Center of Oncological Hadrontherapy (Other)
Responsible Party: Sponsor
Other Study IDs: CNAO OSS 52 2022
Record Dates: First submitted 2023-07-07; First posted 2023-07-17 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Head and Neck Cancer; Skull Base--Cancer; Brain Cancer
Keywords: cancer free survisorship; hadrontherapy; quality of life
MeSH Terms: conditions — Head and Neck Neoplasms; Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cohort A Survivors: about 80 patients with at least a 5 year follow up with head and neck, skull base and brain tumors and no evidence of progressive disease.
  Interventions: Other: questionnaires administration
- Cohort B: 100 patients with histological and/or radiological diagnosis of head and neck tumors enrolled at baseline
  Interventions: Other: questionnaires administration

INTERVENTIONS:
Other: questionnaires administration — Enrolled people will be requested to fill in questionnaires. Cohort A affected by head and neck cancer: SF-12, EORTC QLQ-C30, EORTC QLQ-H&N43, HADS, Brief COPE, BRCS.
  Cohort A affected by skull base/brain cancer: SF-12, EORTC QLQ-BN20, HADS, Brief COPE, BRCS.
  Cohort B will receive: EORTC QLQ-C30, BRCS, PROFFIT, SF-12, EORTC QLQ-H&N43.

SUMMARY:
The Quality of Life of patients treated with hadrontherapy is still limited. Two cohorts are established, they will be receiving specific standardized questionnaires to be evalutaed in their results.

DETAILED DESCRIPTION:
Since 2011, CNAO has been treating patients suffering from solid tumors with particle therapy (both protons and carbon ions). Hadrontherapy improves outcome of radioresistant tumors which normally do not benefit from conventional radiotherapy. The treated population is highly heterogenous in term of tumor site, histotype, treatment fields and doses however its common anatomical origin justifies a unified approach in evaluating a QoL in this setting. QoL of patients suffering from these tumors have been poorly investigated and there are still few studies on patient reported outcomes (PROs) and QoL following hadrontherapy. In this context, therefore, there is a need to generate data by designing distinct cohort studies, conceived within a single protocol, that will gather quality of life data by means of standardized questionnaires of patients along their oncological history. Thanks to this protocol design, the investigator will be facilitated, in the future, in adding new cohorts pending a study protocol amendment and ethical approval.

ELIGIBILITY:
Cohort A ("survivors"):

Inclusion Criteria

* Patients with at least a follow up of 5 years with head and neck, skull base and brain tumors and no evidence of progressive disease.
* The patient is able to give consent

Exclusion Criteria:

* Re-irradiation.
* Second tumor.
* Known cases of any psychiatric and neurological diseases leading to disability (eg, manic disorder, schizophrenia etc..), which could impair compilation of questionnaires or affect quality of life.

Cohort B:

Inclusion Criteria:

* Histological and/or radiological diagnosis of head and neck tumors
* Patients candidate for curative intent hadrontherapy
* Patients ≥ 18 years of age
* The patient is able to give consent

Exclusion criteria:

* Re-irradiation.
* Second tumor
* Known cases of any psychiatric and neurological diseases leading to disability (eg, manic disorder, schizophrenia etc..), which could impair compilation of questionnaires or affect quality of life
* Presence of diffused metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients from cohort A will be selected and invited to participate in the study when evaluated for standard of care follow-up which is taking place in telemedicine modality through a digital meeting organized by the staff.
  Patients from Cohort B with indication of hadrontherapy in radical setting will be consecutively enrolled at baseline (during CT simulation procedure or at the first session of RT).
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2023-03-27 (Actual); Primary Completion 2025-09-26 (Estimated); Study Completion 2025-09-26 (Estimated)

PRIMARY OUTCOMES:
investigate relation between quality of life and several socio- psycho- variables | 5 years follow uo after hadrontherapy
  quality of life in subjects treated with curative hadrontherapy investigated by global score according to Short-form-12-health-survey-questionnaire (SF-12) and compared to healthy population

SECONDARY OUTCOMES:
quality of life related also to psychological variables, socio-cognitive factors, resilience | before treatment and after 1 year from treatment completion
  quality of life in subjects treated with curative hadrontherapy investigated by global score according to EORTC QLQ-C30

CONTACTS AND LOCATIONS:
Overall Officials: Anna Maria Camarda, Principal Investigator — CNAO National Center of Oncological Hadrontherapy
Locations (1):
- CNAO, Pavia, Pv, Italy